CLINICAL TRIAL: NCT01455441
Title: Does the GLP-1 Receptor Agonist (Victoza®) Improve the Metabolic Response to Physical Training in Patients With Type 2 Diabetes?
Brief Title: The Effects of Physical Training and GLP-1 Receptor Agonist Liraglutide Treatment in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tina Vilsboll (Other)
Responsible Party: Sponsor-Investigator, Tina Vilsboll, Professor dr.med, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 60 - TrainIncretin
Record Dates: First submitted 2011-10-19; First posted 2011-10-20 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Type 2 Diabetes
Keywords: GLP-1; Training; Exercise; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Training and liraglutide (Active Comparator): Treatment with both training and liraglutide for 16 weeks
  Interventions: Other: Training and liraglutide
- Training and placebo (Placebo Comparator): Treatment wiht both training and placebo for 16 weeks
  Interventions: Other: Training and placebo

INTERVENTIONS:
Other: Training and liraglutide
  Arms: Training and liraglutide
Other: Training and placebo
  Arms: Training and placebo

SUMMARY:
The objective of this study is to investigate the effects of physical training in patients with type 2 diabetes during treatment with the GLP-1 receptor agonist liraglutide (Victoza®) in a 16-weeks double-blinded, randomized placebo-controlled clinical trial.

Hypothesis: Physical training leads to better metabolic control in type 2 diabetic patients when training is combined with liraglutide (Victoza®) treatment.

ELIGIBILITY:
Inclusion Criteria:

* Informed oral and written consent
* Diagnosed with type 2 diabetes according to the criteria of the WHO
* HbA1C: 7-11% (doing treatment with diet and/or metformin)
* Age >18 years
* BMI >25 kg/m2 <40 kg/m2
* Negative islet cell antibodies (ICA) and glutamate decarboxylase 65 (GAD- 65) autoantibodies

Exclusion Criteria:

* Females of child bearing potential who are pregnant, breast-feeding or have intention of becoming pregnant or are not using adequate contraceptive measures.
* Subjects treated with sulfonylureas, dipeptidyl peptidase 4 (DPP-4) inhibitors, insulin or glitazones
* Ongoing abuse of alcohol or narcotics
* Impaired hepatic function (liver transaminases >2 times upper normal limit)
* Impaired renal function (se-creatinine >150μM and/or albuminuria)
* Cardiac problems defined as decompensated heart failure (NYHA class III or IV), unstable angina pectoris and/or myocardial infarction within the last 12 months
* Uncontrolled hypertension (systolic blood pressure >180 mmHg, diastolic blood pressure >100 mmHg)
* Anaemia
* Any condition that the investigators feels would interfere with trial participation
* Receiving any investigational drug within the last 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-10; Primary Completion 2013-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
HbA1c | 16 weeks
  Change in HbA1c from baseline to 16 weeks. Glycated haemoglobin (HbA1c) is a form of haemoglobin which is measured primarily to identify the average plasma glucose concentration over prolonged periods of time (12 weeks).

SECONDARY OUTCOMES:
Maximal oxygen uptake (VO2peak) | 16 weeks
  Changes in VO2peak from baseline to 16 weeks
Body weight | 16 weeks
  Changes in body weight from baseline to 16 weeks evaluated by a full body DEXA scan
Blood pressure | 16 weeks
  Changes in blood pressure from baseline to 16 weeks
Glycaemic control | 16 weeks
  Changes in overall glycaemic control parameters, insulin sensitivity and beta cell function evaluated by The Homeostasis Model Assessment (HOMA) and incretin hormones response
Meal test | 16 weeks
  The changes in the postprandial response of incretin hormones, insulin and glucose, glucagon and the microvascular blood flow will be evaluated. Changes in blood leves of triglycerides and cholesterol.
Myocardial echocardiography | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Gentofte Hospital, Hellerup, Denmark